CLINICAL TRIAL: NCT02018250
Title: A Phase 1 Double-Blind, Placebo-Controlled, Single-Center Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Intramuscular Administration of a New Oxime, MMB4 DMS Enhanced Formulation (EF)
Brief Title: Study to Evaluate the Safety of a New Oxime, MMB4 DIMETHANESULFONATE (DMS)
Acronym: MMB4(DMS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MMB4-09-1001 S-12-08; S-12-08/A-15399.2 (Other: USAMRMC)
Record Dates: First submitted 2012-12-27; First posted 2013-12-23 (Estimated); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Safety and Efficacy
MeSH Terms: interventions — N,N'-monomethylenebis(pyridiniumaldoxime); Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 0.6 mg/kg MMB4 DMS (Experimental): 0.6 mg/kg 1,1'-Methylenebis[4-[(hydroxyimino) methyl]-pyridinium] dimethanesulfonate (MMB4 DMS), intramuscular (i.m.) to the anterior thigh.
  Interventions: Drug: MMB4 DMS
- Placebo (Placebo Comparator): filtered cottonseed oil for injection. Three and a half milliliter aliquots of the placebo are placed in each 5-mL vial and administered intramuscular (i.m.) to the anterior thigh.
  Interventions: Drug: Placebo
- 0.9 mg/kg MMB4 DMS (Experimental): 0.9 mg/kg 1,1'-Methylenebis[4-[(hydroxyimino) methyl]-pyridinium] dimethanesulfonate (MMB4 DMS), intramuscular (i.m.) to the anterior thigh.
  Interventions: Drug: MMB4 DMS
- 1.2 mg/kg MMB4 DMS (Experimental): 1.2 mg/kg 1,1'-Methylenebis[4-[(hydroxyimino) methyl]-pyridinium] dimethanesulfonate (MMB4 DMS), intramuscular (i.m.) to the anterior thigh.
  Interventions: Drug: MMB4 DMS
- 1.5 mg/kg MMB4 DMS (Experimental): 1.5 mg/kg 1,1'-Methylenebis[4-[(hydroxyimino) methyl]-pyridinium] dimethanesulfonate (MMB4 DMS), intramuscular (i.m.) to the anterior thigh.
  Interventions: Drug: MMB4 DMS

INTERVENTIONS:
Drug: MMB4 DMS — Subjects will be administered the drug product formulation at the assigned dosage of MMB4 DMS or placebo i.m. to the anterior thigh using a 5 mL syringe.
  Other Names: 1,1'-methylenebis[4-[(hydroxyimino)methyl]-pyridinium] dimethanesulfonate
  Arms: 0.6 mg/kg MMB4 DMS; 0.9 mg/kg MMB4 DMS; 1.2 mg/kg MMB4 DMS; 1.5 mg/kg MMB4 DMS
Drug: Placebo — Subjects will be administered the drug product formulation at the assigned dosage of placebo i.m. to the anterior thigh using a 5 mL syringe. The placebo group in each cohort will receive the same injection volume and number of injections as the dose group in that cohort.
  Other Names: Benzyl alcohol USP/NF and methanesulfonic acid adjusted to a pH 2.3
  Arms: Placebo

SUMMARY:
This clinical study will evaluate escalating dosages of MMB4 DMS to determine its safety when delivered intramuscularly (i.m.) to the anterior thigh.

DETAILED DESCRIPTION:
The goal of this study is to assess safety, tolerability, and PK of MMB4 DMS EF at up to six cohorts chosen to provide the range required for PK analyses, including assessment of dose proportionality.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be generally healthy adult male or female volunteers, 18-to-55 years-of age;
* Subjects must be physically fit as determined by physical examination and BMI;
* Subjects must have BMI of ≥ 19 and ≤ 30 kg/m2, and weight range of 55-85 kg;
* Subjects must have adequate venous access;
* Females of child bearing age must not be pregnant or breast-feeding, nor plan to become pregnant for the duration of the study, and all females must have a negative serum pregnancy test within 28 days of treatment, and a negative serum pregnancy test prior to dosing;
* Females of childbearing potential must have been using adequate contraception, defined as the use of hormonal (oral, injectable, or implantable) or barrier-method contraceptives for at least one month prior to drug administration and must agree to use an adequate method of contraception for at least one month following drug administration. Women who are lactating will be excluded. Women without childbearing potential (who have undergone a total hysterectomy or bilateral oophorectomy, have a history of bilateral tubal ligation, or are two years post-menopausal) are also eligible;
* Males must agree to use a barrier form of birth control (i.e., condom with spermicidal gel) from the time of check-in to the clinical unit to 30 days after exposure to the study drug;
* In the opinion of the Investigator, subjects who comply with the protocol and are likely to complete the study;
* Subjects must provide written informed consent by signing and dating an IRB-approved written informed consent before any screening procedures are performed;
* Subjects must be willing to refrain from donating blood for eight weeks after completion of the study period;
* Subjects must be able to read/comprehend English; and
* Subjects are non-smokers/tobacco/nicotine product users within three months of first dosing and must have a total lifetime exposure to cigarettes of <15 pack-years.

Exclusion Criteria:

* Participation in a PK study or any other clinical study currently or within the last 30 days;
* History or presence of significant cardiovascular, hepatic, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease that could potentially impact the safety of the subject or metabolism of the drug;
* Have an active malignancy or history of metastatic or hematologic malignancy with the exception of melanoma in situ or basal or squamous cell carcinoma of the skin. Subjects must be disease-free for ten years;
* History of glaucoma;
* History of seizures;
* History of allergic or untoward reaction to any bispyridinium oximes; or history allergy to cotton seed oil or history of anaphylactic shock;
* History of chronic pulmonary disease or current acute pulmonary disease; history of treatment for asthma or any other reactive airways disease in the past year;
* Have ongoing drug abuse/dependence (including alcohol); or recent history (over the past five years) of treatment for alcohol or drug abuse; or a current positive urine tests for drug abuse;
* Have consumed grapefruit, grapefruit juice, other grapefruit containing products, or starfruit within seven days prior to planned dosing;
* Having taken, within 14 days of planned dosing, any prescription or non-prescription medication (including home remedies, herbal supplements or nutritional supplements) unless the Principal Investigator/Sub-Investigator, in consultation with the Sponsor Medical Monitor, provides a statement justifying that the medication taken will not impact the results of this study (with rare exceptions taking prescriptions drugs will be grounds for exclusion);
* Preexistent renal insufficiency (estimated GFR using a GFR prediction equation <60 mL/min/1.73m^2, and/or other evidence of structural or functional abnormalities (e.g. PI assessment of the presence of clinically significant hematuria, proteinuria, or history of abnormalities on renal imaging) and/or abnormal BUN and serum creatinine or an abnormal urinalysis;
* Skeletal muscle disease or evidence of skeletal muscle injury based on abnormal (>1.5 x ULN) blood creatine kinase and myoglobin levels;
* Clinically relevant abnormal physical findings (including vital signs, pulse oximetry, and transcutaneous or end-tidal PCO2) or laboratory values at the pre-study period screening assessment that could interfere with the objectives of the study or the safety of the subject;
* Clinically relevant ECG abnormalities based on three 12-lead ECGs obtained five minutes apart;
* ECG with a PR interval ≥ 200 msec at screening or before dosing;
* ECG with a QTc interval > 450 msec for males, 470 msec for females (QT interval corrected with Bazett formula);
* Supine blood pressure less than 100/55 mmHg at screening or before dosing;
* Ejection fraction less than 55% on screening echocardiogram;
* Have spirometry with abnormal FEV1, FVC or FEV1/FVC ratio according to current American Thoracic Society/European Respiratory Society standards.
* Have any specified laboratory values (e.g., hematology - complete blood count with differential, serum chemistry and urinalysis) outside the normal range for age and sex and deemed clinically significant by the Principal Investigator, within 28 days before treatment;
* Have positive tests for hepatitis B surface antigen, hepatitis C, syphilis, human immunodeficiency virus (HIV) HIV-1 or HIV-2;
* Have any skin condition that would interfere with injection of study drug; or
* Donated >480 mL of blood in the last 8 weeks.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-03-17 (Actual); Primary Completion 2012-10-16 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events (AE) | 30 days post-administration

SECONDARY OUTCOMES:
Safety electrocardiogram (ECG) (3-5 lead) | Up to 48-hours post administration
Oxygen saturation | Up to 48-hours post administration
End-Tidal carbon dioxide | Up to 48 hours post administration
Blood pressure | Up to 48 hours post administration

OTHER OUTCOMES:
Observed Cmax | Multiple timepoints between 0 and 24 hours
  Samples will be analyzed for MMB4 using a validated high performance liquid chromatography-tandem mass spectrometry (HPLC/MS/MS)
Observed Tmax | Multiple timepoints between 0 and 24 hours
  Samples will be analyzed for MMB4 using a validated high performance liquid chromatography-tandem mass spectrometry (HPLC/MS/MS). Samples will be evaluated using semi-log plots and characterized using non-compartmental analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S Al-Ibrahim, MD, Principal Investigator — SNBL Clinical Pharmacology Center, Inc.
Locations (1):
- SNBL Clinical Pharmacology Center, Inc., Baltimore, Maryland, United States